CLINICAL TRIAL: NCT02398591
Title: A Double-blind, Placebo-controlled, Randomized, Single Ascending Dose Study to Investigate Safety, Tolerability, and Pharmacokinetics of JNJ 53718678 in Healthy Japanese Adult Subjects
Brief Title: A Study to Investigate Safety, Tolerability, and Pharmacokinetics of JNJ 53718678 in Healthy Japanese Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Sciences Ireland UC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR107003; 53718678RSV1004 (Other: Janssen Sciences Ireland UC); 2014-005410-36 (EudraCT Number)
Record Dates: First submitted 2015-03-20; First posted 2015-03-25 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Healthy
Keywords: Healthy; JNJ 53718678
MeSH Terms: interventions — JNJ-53718678

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (3):
- JNJ 53718678 250 milligram (mg) (Experimental): Participants will receive either single oral dose of 250 mg of JNJ 53718678 or matching placebo on Day 1.
  Interventions: Drug: JNJ 53718678; Drug: Placebo
- JNJ 53718678 500 mg (Experimental): Participants will receive either single oral dose of 500 mg of JNJ 53718678 or matching placebo on Day 1.
  Interventions: Drug: JNJ 53718678; Drug: Placebo
- JNJ 53718678 1000 mg (Experimental): Participants will receive either single oral dose of 1000 mg of JNJ 53718678 or matching placebo on Day 1.
  Interventions: Drug: JNJ 53718678; Drug: Placebo

INTERVENTIONS:
Drug: JNJ 53718678 — JNJ 53718678 will be orally administered once in a dose of 250, 500 or 1000 mg on Day 1.
Drug: Placebo — Placebo matching to JNJ 53718678 will be orally administered once on Day 1.

SUMMARY:
The purpose of this study is to investigate the safety, tolerability, and pharmacokinetics of three dosages (250, 500, and 1000 milligram [mg], or maximum tolerated dose [MTD]) of JNJ 53718678 when administered as single dose in fasting conditions in healthy Japanese adult participants in 3 cohorts.

DETAILED DESCRIPTION:
This is a Phase 1, single center, double-blind (study in which neither the researchers nor the participants know what treatment the participants are receiving), placebo-controlled (study in which the experimental treatment or procedure is compared to placebo treatment), randomized (study medication assigned to participants by chance) study in healthy Japanese adult participants residing outside of Japan. The study will consist of a Screening phase, an In-clinic treatment phase, and a follow-up phase. The study duration for each participant will be approximately 6 weeks from Screening (Day -28 to Day -2) to follow up visit (Day 10 to 14). Participants will be randomly assign to receive JNJ 53718678 or placebo, at planned dose of 250, 500 and 1000 milligram (mg). Planned doses will be stepwise escalated, if the safety and tolerability of the preceding dose(s) are found to be acceptable, and the maximum tolerated dose (MTD) is not reached. De-escalation may be performed in order to study an intermediate dose. The safety, tolerability and pharmacokinetic (PK) profile of JNJ-53718678 will primarily be evaluated. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be a Japanese participant who has resided outside Japan for no more than 5 years and whose parents and grandparents are Japanese as determined by participant's verbal report
* Participant must be healthy on the basis of a medical evaluation that reveals the absence of any clinically relevant abnormality and includes a physical examination (including height and body weight measurement and skin examination), medical history, vital signs (body temperature, systolic blood pressure, diastolic blood pressure, pulse rate, orthostatic hypotension, and respiratory rate), and the results of blood biochemistry, blood coagulation and hematology tests, a urinalysis, and a hematest performed at Screening, on Day -1, or Day 1 pre-dose, whichever is applicable. If there are abnormalities, the participant may be included only if the Investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the Investigator
* Female participants must be of non-childbearing potential: postmenopausal for at least 2 years (amenorrheal for at least 2 years and a serum follicle stimulating hormone [FSH] level greater than [>] 40 international unit per liter [IU/L] or milli IU per milliliter [mIU/mL]), or surgically sterile (have had a total hysterectomy, bilateral oophorectomy, or bilateral tubal ligation/bilateral tubal clips without reversal operation), or otherwise incapable of becoming pregnant
* Participant must be a non-smoker for at least one month prior to Screening
* Participant must have a body mass index (BMI) (weight [kilogram{kg}]/height^2 [meter^2]) between 18 and 30 kg/m^2 (inclusive), and body weight not less than 50 kg

Exclusion Criteria:

* Participant has a history of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the Investigator considers should exclude the subject or that could interfere with the interpretation of the study results
* Participant with any history of clinically significant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, and urticaria
* Clinically significant abnormal physical examination, vital signs, or 12 lead electrocardiogram (ECG) at Screening, on Day -1 (physical examination only), and pre-dose on Day 1, as deemed appropriate by the Investigator
* Participants with lack of good/reasonable venous access
* Participants with a past history of heart arrhythmias (extrasystoli, tachycardia at rest) or, history of risk factors for Torsade de Pointes syndrome (for example, hypokalemia, family history of long QT Syndrome

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2015-07-15 (Actual); Study Completion 2015-07-15 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Up to 72 hours post dose
  The Cmax is the maximum observed plasma concentration.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Up to 72 hours post dose
  The Tmax is defined as actual sampling time to reach maximum observed JNJ 53718678 concentration.
Time to Last Quantifiable Plasma Concentration (Tlast) | Up to 72 hours post dose
  The Tlast is the time to last observed quantifiable plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) | Up to 72 hours post dose
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) | Up to 72 hours post dose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Apparent Initial Elimination Rate Constant (lambda [alpha]) | Up to 72 hours post dose
  Apparent initial elimination rate constant, determined by linear regression of the data points within the first elimination phase of the ln-linear plasma concentration-time curve.
Elimination Rate Constant (Lambda[z]) | Up to 72 hours post dose
  Lambda(z) is first-order elimination rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Apparent Initial Elimination Half-life (t1/2[alpha]) | Up to 72 hours post dose
  Apparent initial elimination half-life is calculated as 0.693/lambda(alpha).
Elimination Half-Life (t1/2) | Up to 72 hours post dose
  The elimination half-life (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Total Apparent Clearance (CL/F) | Up to 72 hours post dose
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vd/F) | Up to 72 hours post dose
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after subcutaneous dose (Vd/F) is influenced by the fraction absorbed.
Number of Participants With Adverse Events | From sign of informed consent up to end of study (Day 14)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Sciences Ireland UC Clinical Trials, Study Director — Janssen Sciences Ireland UC
Locations (1):
- Harrow, United Kingdom